CLINICAL TRIAL: NCT05657197
Title: ENERGIZE IBD - The Effect of Intensive Physical Exercise on Fatigue and Quality of Life in Patients With Quiescent Inflammatory Bowel Disease: A Randomized Controlled Trial
Brief Title: The Effect of Intensive Physical Exercise on Fatigue and Quality of Life in Patients With Quiescent Inflammatory Bowel Disease
Acronym: ENERGIZE-IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: Dutch Digestive Diseases Foundation (Other); Sport Medisch Centrum Papendal (Unknown); FormUpgrade, Arnhem (Unknown); Sport Medisch Centrum, Jeroen Bosch Ziekenhuis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL81794.091.22
Record Dates: First submitted 2022-10-24; First posted 2022-12-20 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Fatigue; Exercise; Quality of life; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fatigue; Motor Activity

STUDY DESIGN:
Masking Description: Multicentre parallel randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (exercise) group (Experimental): The patients in the intervention group will follow a personalised and intensive exercise program.
  Interventions: Behavioral: Exercise intervention
- Control group (Other): The patients in the control group will receive usual care.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Exercise intervention — A 12-week exercise program consisting of three times per week 1-hour sessions, including 30-minutes aerobic- and 30-minutes progressive resistance training. The intensity of training will be adjusted to each individual, based on a cardiopulmonary exercise test. Training sessions will be performed in groups of 10 participants under supervision of a sports physical therapist.
  Arms: Intervention (exercise) group
Other: Usual care — Usual care, including general advice concerning chronic fatigue.
  Arms: Control group

SUMMARY:
In patients with inflammatory bowel diseases (IBD), characterized by relapsing intestinal inflammation, chronic fatigue is a burdensome and highly prevalent symptom. The aetiology is thought to be multifactorial, including complex interactions of psychological and physical factors such as immunological profiles and gut microbiota. Unfortunately, specific treatment strategies are currently lacking. Since fatigued patients have an impaired physical fitness and are less physically active than patients without fatigue, it is hypothesised that physical exercise might be an effective complementary treatment for patients with IBD suffering from fatigue. During a previous pilot cohort study, significant improvements in fatigue complaints and quality of life were observed following a personalised and intensive exercise program. In this study, a multicenter randomized controlled trial will be performed to further investigate this assumed beneficial effect of intensive physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 year diagnosis of IBD, including Crohn's disease (CD), ulcerative colitis (UC) and IBD-unclassified (IBD-U), based on a combination of clinical, endoscopic, histologic and radiologic internationally accepted criteria;
* Chronic fatigue complaints for at least 3 months;
* Severe fatigue complaints as confirmed with a score of ≥11 on section I of the inflammatory bowel disease fatigue self-assessment scale (IBD-F);
* Clinically quiescent IBD with a Harvey Bradshaw Index (HBI) <5 for Crohn's disease patients or a Simple Colitis Clinical Activity Index (SCCAI) ≤2 for patients with ulcerative colitis or IBD-unclassified;
* Faecal calprotectin <100 μg/g;
* Stable medication for at least 3 months before screening visit;
* Patient is able and willing to provide written informed consent;
* Patient is able/commitment to make a time investment to complete the intervention program (one hour training 3x/week during 12 weeks) or, after randomisation, willing to participate in the control group;
* Patient is aged between 18 and 60 years.

Exclusion Criteria:

* Performing moderate-vigorous intensity exercise (i.e. swimming, running, cycling) more than once and/or >90 minutes per week in the past 3 months;
* Surgery within the past 6 months or planned surgery within 12 months after the screening visit;
* Participation in another intervention study;
* Pregnant at the moment of the screening visit or planning pregnancy within 12 months after the screening;
* Confirmed diagnosis of other causes of fatigue complaints, such as thyroid dysfunction, liver or renal failure, anaemia, folate-, iron-, vitamin B12- or D deficiency.
* Comorbidities that could be confounders for fatigue, such as Chronic obstructive pulmonary disease (COPD), heart failure, active malignancy, long/Post-COVID and patients under treatment for a psychiatric disorder (i.e. depression/anxiety)
* Comorbidities that prevent safe participation in the exercise program/cardiorespiratory fitness test including;

  * Very high risk of cardiovascular disease
  * Uncontrolled diabetes mellitus with HbA1c > 65 mmol/l.
  * Cardiovascular disease (i.e. acute myocardial infarct, unstable angina, uncontrolled arrhythmias, aortic stenosis, stenotic valvular heart disease, untreated arterial hypertension (>200 mmHg systolic, >120 mmHg diastolic))
  * Acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise (i.e. infection, thyrotoxicosis)
  * Uncontrolled asthma
  * Pulmonary oedema
  * Significant pulmonary hypertension
  * Acute pulmonary embolus or pulmonary infarction
  * Room air desaturation at rest <85% (exercise with supplemental O2)
  * Respiratory failure
  * Electrolyte abnormalities (sodium, potassium, calcium, magnesium)
  * Mental impairment leading to inability to cooperate
  * Orthopaedic impairment that compromise exercise performance
  * BMI ≥35

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue (IBD-F), post-intervention | 3 months (post-intervention)
  Mean change in fatigue, measured with the inflammatory bowel disease fatigue self-assessment scale (IBD-F) 0-140 with higher scores indicating worse fatigue, in the intervention group compared to the control group.
Change in quality of life (IBDQ), post-intervention | 3 months (post-intervention)
  Mean change in quality of life, measured with the inflammatory bowel disease questionnaire (IBDQ) 32-224 with higher scores representing better quality of life, in the intervention group compared to the control group.

SECONDARY OUTCOMES:
Long-term change in fatigue (IBD-F) | 6- and 12-months
  Mean change in fatigue, as measured after 6- and 12-months using the IBD-F, in the intervention group compared to the control group
Long-term change in quality of life (IBDQ) | 6- and 12-months
  Mean change in quality of life, as measured after 6- and 12-months using the IBDQ, in the intervention group compared to the control group
Change in cardiorespiratory fitness (maximum oxygen uptake) | 3 months (post-intervention)
  Change in cardiorespiratory fitness (maximum oxygen uptake) of patients in the intervention group, assessed using Cardiopulmonary Exercise Testing (CPET).
Change in cardiorespiratory fitness (maximum power) | 3 months (post-intervention)
  Change in cardiorespiratory fitness (maximum power) of patients in the intervention group, assessed using Cardiopulmonary Exercise Testing (CPET).
Change in muscular strength | 3 months (post-intervention)
  Change in muscular strength of patients in the intervention group, assessed using one-repetition maximum (1-RM)
Change in body composition (BMI) | 3 months (post-intervention)
  Change in body composition in the intervention group, as determined by body mass index (BMI).
Change in body composition (body fat percentage) | 3 months (post-intervention)
  Change in body composition in the intervention group, as determined by body fat percentage measured using skinfold techniques
Change in work absenteeism and presenteeism | T= 3-, 6-, 9-, and 12-months
  Change in work absenteeism and presenteeism in the intervention group compared to the control group, as measured by the Productivity Cost Questionnaire (iPCQ)
Disease activity (FCP) | T= 3-, 6-, 9-, and 12-months
  Disease activity measured by change in faecal calprotectin (FCP), in both the intervention- and control group
Disease activity (step-up therapy) | T= 3-, 6-, 9-, and 12-months
  Disease activity measured by step-up therapy rate in both the intervention- and control group
Disease activity (exacerbation rate) | T= 3-, 6-, 9-, and 12-months
  Disease activity measured by exacerbation rate in both the intervention- and control group
Change in sleep quality | T= 3-, 6-, 9-, and 12-months
  Self-reported differences in sleep quality in the intervention group compared to the control group, using the Pittsburgh Sleep Quality Index (PSQI), 0-21 with higher scores indicating worse sleep quality.
Change in anxiety and depression symptoms | T= 3-, 6-, 9-, and 12-months
  Mean change in anxiety and depression symptoms in the intervention group compared to the control group, measured using the Hospital Anxiety and Depression Scale (HADS) questionnaire, each subscale 0-21 higher scores indicating worse symptoms
Targeted cost-utility analysis | 12 months
  Targeted economic evaluation of the intervention using a targeted cost-utility analysis from a societal perspective including intervention costs, medical consumption costs and productivity loss. Effectiveness of the intervention will be determined using the mean Difference of quality adjusted life years (QALYs) between de intervention and control group, based on the designated EQ-5D-5L questionnaire.
Exploratory outcome measurements (immunological profiles) | 3 months (post-intervention)
  Differences in the immunological profiles (i.e. pro- and anti-inflammatory cytokines and soluble receptors, such as IL-10, IL-6, IFN-ɣ) in the intervention group compared to the control group
Exploratory outcome measurements (gut microbiota) | 3 months (post-intervention)
  Differences in the gut microbiota diversity and composition in the intervention group compared to the control group using 16SrRNA sequencing.
Exploratory outcome measurements (biogenic amines) | 3 months (post-intervention)
  Differences in the concentration of biogenic amines in the intervention group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. M.J.M. Groenen, MD, PhD, Principal Investigator — Gastroenterology department, Rijnstate Hospital
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Radboud Univeristy Medical Center, Nijmegen, Gelderland
  - Jeroen Bosch Hospital, 's-Hertogenbosch, S' Hertogenbosch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Erp LW, Roosenboom B, Komdeur P, Dijkstra-Heida W, Wisse J, Horjus Talabur Horje CS, Liem CS, van Cingel REH, Wahab PJ, Groenen MJM. Improvement of Fatigue and Quality of Life in Patients with Quiescent Inflammatory Bowel Disease Following a Personalized Exercise Program. Dig Dis Sci. 2021 Feb;66(2):597-604. doi: 10.1007/s10620-020-06222-5. Epub 2020 Apr 1. PMID 32239380